CLINICAL TRIAL: NCT02448472
Title: Chinese Epidemiological Study of Severe Sepsis.(CHESS Study)
Brief Title: Epidemiology of Sepsis in China
Status: Completed | Type: Observational
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, Attending, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: 20150315
Record Dates: First submitted 2015-04-11; First posted 2015-05-19 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2015-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Observational study, none intervention

SUMMARY:
Sepsis is a common cause for morbidity and mortality in critically ill patients. In USA, the incidence of sepsis is about 3/1000 population. However, the incidence of sepsis varies among different clinic trails. In addition, clinician empirical select antibiotic according to the epidemiology of sepsis, however, the etiology of sepsis is various in different studies. In China, the MDRO is much higher than western country. There is no study about the epidemiology of sepsis in China. Therefore, it is necessary to conduct a study about it in China.

DETAILED DESCRIPTION:
Sepsis,especially severe sepsis is a major cause of admission to the intensive care unit (ICU) and death. In USA, the incidence of sepsis is about 3/1000 population. However, the incidence of sepsis varies among different clinic trails. Between 6 and 54% of patients admitted to ICUs have severe sepsis and the mortality rate for these patients varies from 20 to 60%. There is no exactly results of incidence of sepsis in China.

In addition, clinician empirical select antibiotic according to the epidemiology of sepsis, however, the etiology of sepsis is various in different studies. In EPIC II study, the organisms of sepsis include Gram-positive microorganisms (69.8%),Gram-negative microorganisms(62.2%) and fungi (17%). In China, the MDRO is much higher than western country. In contrast to EPIC II study, one study in China showed that the organisms of sepsis include Gram-positive microorganisms (14.5%),Gram-negative microorganisms(62.5%) and fungi (2.2%). Therefore, it is necessary to conduct a study about epidemiology of sepsis in China.

ELIGIBILITY:
Inclusion Criteria:

sepsis patients who admitted into ICU during research period (include patients with sepsis at ICU admission and patients who has new sepsis during ICU period)

Exclusion Criteria:

The patients with second sepsis in ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sepsis patient who admitted into ICU
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence | Patients will be assessed up to 90 days
Mortality | Sepsis and severe sepsis patients will be assessed up to 90 days

SECONDARY OUTCOMES:
etiology | The pathogen of sepsis will be assessed up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yi, Ph.D., Study Director — Zhongda Hospital
Locations (1):
- Zhongda hospital, Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Xie J, Wang H, Kang Y, Zhou L, Liu Z, Qin B, Ma X, Cao X, Chen D, Lu W, Yao C, Yu K, Yao X, Shang H, Qiu H, Yang Y; CHinese Epidemiological Study of Sepsis (CHESS) Study Investigators. The Epidemiology of Sepsis in Chinese ICUs: A National Cross-Sectional Survey. Crit Care Med. 2020 Mar;48(3):e209-e218. doi: 10.1097/CCM.0000000000004155. PMID 31804299
- [Derived] Yang Y, Xie JF, Yu KJ, Yao C, Li JG, Guan XD, Yan J, Ma XC, Kang Y, Yang CS, Yao XQ, Shang HC, Qiu HB; for CHESS Study Investigators. Epidemiological Study of Sepsis in China: Protocol of a Cross-sectional Survey. Chin Med J (Engl). 2016 Dec 20;129(24):2967-2973. doi: 10.4103/0366-6999.195474. PMID 27958229